CLINICAL TRIAL: NCT07074197
Title: The Effect of Smelling the Scent of Infants Hospitalized in the Neonatal Intensive Care Unit on Mothers' Stress, Attachment and Perception of Insufficient Milk
Brief Title: The Effect of Smelling the Scent of Infants Hospitalized in the Neonatal Intensive Care Unit
Acronym: NICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Dilek Kucuk Alemdar, Professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KAEK86
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: NICU
Keywords: NICU; infant; mother; stress; scent; attachment

STUDY DESIGN:
Intervention Model Description: The study was a randomized controlled experimental, prospective study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: After the mothers of newborns who met the inclusion criteria were randomly assigned to the study groups, written informed consent was obtained without informing the parents about which group their infants would be included in. The researcher placed the OOKIE baby next to the infant herself and then gave it to the mother, so the researcher was not blinded. However, to avoid bias, the outcome measures were recorded by two nurses working in the NICU, who were university graduates and did not know which mother was in the experimental or control group. To avoid bias during data analysis, the database of the study groups was coded as A and B by someone other than the researcher, and the data were analyzed by an independent statistician. Blinding of outcome measurements, statistical analysis and reporting was performed to prevent statistical and reporting bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control group: No intervention was made except for the routine care provided at the clinic where the study was conducted. Routine practices included allowing the mother to visit and see her baby at the clinic whenever she wanted. When the mother came for the first visit, the mother and baby introductory information form, Neonatal Intensive Care Unit Parent Stress Scale, Inadequate Milk Perception Scale, Mother-Infant Attachment Scale and NICU Parental Beliefs Scale pretest were administered. On the third day, when the mothers came to visit their babies, the same scales were administered as posttest.
- OOKİE group (Experimental): The infants who met the selection criteria were wrapped with OOKIE upon admission and remained in contact with OOKIE for approximately 24 hours without affecting their routine care and position. After 24 hours, when the mother came for the first visit, the mother and baby introductory information form, Neonatal Intensive Care Unit Parent Stress Scale, Inadequate Milk Perception Scale, Mother-Infant Attachment Scale and NICU Parental Beliefs Scale pretest were administered. During the visit, the mother received the OOKIE wrapped around her baby in the incubator and stayed with the mother for 3 days and the mother could smell her baby's odor whenever she wanted.
  The OOKIE used in the study is a doll made of 100% cotton flannel fabric, with satin edges, 35cmx 40cm in size and produced in various colors. Due to its structure, it can be easily washed, dried and sterilized. The fabric feature is capable of trapping and transferring odor. It is a suitable tool for mothers who are separated
  Interventions: Other: OOKIE doll

INTERVENTIONS:
Other: OOKIE doll — The infants who met the selection criteria were wrapped with OOCIE upon admission and remained in contact with OOCIE for approximately 24 hours without affecting their routine care and position. After 24 hours, when the mother came for the first visit, the mother and baby introductory information form, Neonatal Intensive Care Unit Parent Stress Scale, Inadequate Milk Perception Scale, Mother-Infant Attachment Scale and NICU Parental Beliefs Scale pretest were administered. During the visit, the mother received the OOKIE wrapped around her baby in the incubator and stayed with the mother for 3 days and the mother could smell her baby's odor whenever she wanted.
  Arms: OOKİE group

SUMMARY:
The study was conducted to determine the effect of having mothers with infants in the neonatal intensive care unit smell their baby's odor with OOKIE dolls on stress, attachment and perception of insufficient milk.

DETAILED DESCRIPTION:
The infant who met the study selection criteria was wrapped with OOCIE upon admission and remained in contact with OOCIE for approximately 24 hours without affecting routine care and positioning. After 24 hours, when the mother came for the first visit, the mother and baby introductory information form, Neonatal Intensive Care Unit Parent Stress Scale, Inadequate Milk Perception Scale, Mother-Infant Attachment Scale and NICU Parental Beliefs Scale pretest were administered. During the visit, the mother took the OOKIE wrapped around her baby in the incubator and stayed with the mother for 3 days and the mother could smell her baby's odor whenever she wanted.

OOKIE, which will be used in the study, is a doll made of 100% cotton flannel fabric, with satin edges, 35cmx 40cm in size and produced in various colors. Due to its structure, it can be easily washed, dried and sterilized. The fabric feature is capable of trapping and transferring odor. It is a suitable tool for mothers who are separated from their babies in the intensive care environment, which can mediate the smell of their babies.

ELIGIBILITY:
Inclusion Criteria:

* The mother's voluntary acceptance to participate in the study.
* The baby received treatment for at least 3 days in the NICU,
* The baby did not have any congenital anomaly, and the baby did not undergo any surgical procedure.

Exclusion Criteria:

* Mother's illiteracy,
* Mother's having an obstacle to communication,
* Referral of the baby to another center,
* Mother's having an obstacle to breastfeeding or mothers who do not want to breastfeed,
* Mother's having an olfactory problem.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 60 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Neonatal Intensive Care Parent Stress Scale | 1-4. day
  Parents were asked to rate the level of stress caused by each of the factors in the scale from one (no stressor) to five (extreme stressor). Factors with a mean score between 3.0 and 3.40 are considered moderately stressful, and factors with a mean score >3.40 are considered very stressful. Stress factors are analyzed in 3 subgroups. The first is the "Sights and Sounds" subgroup, which includes factors such as the presence of equipment on the baby or in the intensive care unit, sounds arising from them and the environment. The second is the "Appearance and Behavior of the Baby" subgroup, and the third is the factors related to the "Role of the Parents". While filling in the statements such as the presence of tubes and other equipment on or near the baby, sudden change in the baby's color or the baby's breathing stopping, mothers whose babies did not have these symptoms did not mark these items.
Inadequate Milk Perception Scale | 1-4. day
  The inadequate milk perception scale is a form consisting of 6 questions. In the first question, the mother is asked whether she believes that she is feeding her baby enough. The mother answers this question as "yes" or "no". The other questions of the scale aim to measure the perception of milk insufficiency. The mother is asked to score these questions between 0-10. "0" indicates that milk is perceived as completely inadequate and "10" indicates that milk is perceived as completely adequate. A minimum score of 0 and a maximum score of 50 can be obtained from the scale. A higher total score indicates a higher perception of milk adequacy. In the original scale, Cronbach α value was determined as 0.81.
Mother-Infant Attachment Scale | 1-4.day
  The scale is designed to be applied from the first day after birth and allows the mother to express her feelings towards her baby with a single word. The Mother-Infant Attachment Scale (MICS) is a 4-point Likert scale consisting of 8 items. The responses consisting of four options are scored between 0-3, with the lowest score being 0 and the highest score being 24. In the evaluation, items 1, 4, and 6 are positive emotion expressions and are scored as 0,1,2,3, while items 2, 3, 5, 7, and 8 are negative emotion expressions and are scored as 3,2,1,0.
NICU Parental Beliefs Scale | 1-4.day
  The scale is a 5-point Likert-type scale consisting of a total of 18 items. Each item is scored from 1 (strongly disagree) to 5 (strongly agree). The highest score that can be obtained from the scale is 90 and the lowest score is 18. The scale has three sub-dimensions: Parental Role Confidence, Parent-Baby Interaction and Knowledge of the NICU. Higher scores indicate higher parental beliefs and lower scores indicate lower parental beliefs.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Küçük Alemdar, professor, Study Director — Ordu University
Locations (1):
- Ordu University, Altinordu, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No